CLINICAL TRIAL: NCT03892850
Title: Effectiveness and Safety of the Nursing Prescription in Acute Health Problems of Low Complexity. Randomized Clinical Trial
Brief Title: Effectiveness and Safety of the Nursing Prescription in Acute Health Problems of Low Complexity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4R18/112
Record Dates: First submitted 2019-03-18; First posted 2019-03-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Acute Disease
Keywords: Prescriptions; Nurses; Primary Health Care; Acute Disease
MeSH Terms: conditions — Acute Disease | interventions — Prescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nurse prescription (Experimental): experimental group receiving pharmacological nurse prescription
  Interventions: Behavioral: Nurse prescription
- medical prescription (Active Comparator): control group receiving medical prescription
  Interventions: Behavioral: Medical prescription

INTERVENTIONS:
Behavioral: Nurse prescription — Pharmacological nurse prescription. Subjects are individuals who request a same day consultation for minor acute pathologies and meet the selection criteria
  Arms: nurse prescription
Behavioral: Medical prescription — Pharmacological medical prescription. Subjects are individuals who request a same day consultation for minor acute pathologies and meet the selection criteria
  Arms: medical prescription

SUMMARY:
Objective: To compare the efficacy/effectiveness of pharmacological nurse prescription with medical prescription in patients attended in a primary care center for minor acute health problems.

Scope of the study: Multicenter study, with the participation of 8 primary care centers of Catalonia.

Methodology: Randomized blind clinical trial, with experimental group receiving pharmacological nurse prescription and a control group receiving medical prescription. Subjects are individuals who request a same day consultation for minor acute pathologies and meet the selection criteria, with random assignment of 374 subjects, 187 per group.

The efficacy/effectiveness of the prescribed treatment will be considered as a no re-attendance during the following 72h and will be completed with the variables: information and knowledge of the treatment, adverse effects, compliance, satisfaction level and resolution of the health problem. The data collection is done 10 days after the visit by an ad-hoc telephone questionnaire of 11 items, previously tested. The analysis is done using the SPSS software version 21.0, obtaining data of descriptive, multivariate and inferential statistics.

Implications for practice: To evidence the equivalence of pharmacological nurse prescription with medical prescription for minor acute health problems

ELIGIBILITY:
Inclusion Criteria:

* Contusion
* Diarrhea / vomit
* Fever without focality
* Flu
* Urinary distress
* Odinophagy
* Toothache
* Skin Bite
* Upper respiratory symptoms
* Ankle twist

Exclusion Criteria:

* Language barrier
* Cognitive deterioration
* Sensory deficit
* Pregnancy
* Immunosuppression
* Neoplasia in the last 5 years
* Does not participate / Does not sign consent
* Breastfeeding period
* Reconsult
* Resides outside of Spain
* Treatment with glucocorticoids in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
no re-attendance during the following 72 hours | During next 72 hours
  Options: Yes / No

SECONDARY OUTCOMES:
Level of information and knowledge of the treatment | after 10 days
adverse effects | after 10 days
satisfaction level | after 10 days
  Options of survey: Very satisfied, satisfied, ok, dissatisfied, very dissatisfied
resolution of the health problem | after 10 days
  Options of survey: Fully resolved, Very resolved, Something solved, A little resolved, Nothing solved
compliance | after 10 days
  Options: Yes / No (Reason for answered no: Appearance of side effects, Disappearance of symptoms, Distrust of tto, Complicated dosage, No improvement of symptoms, I forget)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Fernandez Molero, Sonia, Principal Investigator — Institut Universitari d'Investigació en Atenció Primària IDIAP Jordi Gol

IPD SHARING:
Plan to Share IPD: No